CLINICAL TRIAL: NCT00466830
Title: Study of Psychological and Sociological Predisposing the Development of Chronic Pain After Surgery in Women With Resectable Breast Cancer
Brief Title: Psychological and Social Factors and Risk Chronic Pain After Surgery in Women With Breast Cancer
Acronym: SDPM
Status: Withdrawn | Type: Observational
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Other Study IDs: IB-2005-31
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Pain; Psychosocial Effects of Cancer and Its Treatment
Keywords: pain; psychosocial effects of cancer and its treatment; stage IIIA breast cancer; stage IIIB breast cancer; stage I breast cancer; stage II breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionnaire administration
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
Certain psychological and social factors may increase the risk of developing chronic pain after surgery. Evaluating these factors over time in patients who have undergone surgery for breast cancer may help doctors plan treatment and improve patients' quality of life.

This clinical trial is studying the psychological and social factors that may increase the risk of developing chronic pain after surgery in women with breast cancer .

DETAILED DESCRIPTION:
OBJECTIVES:

Primary : Determine the psychological and sociological factors that predispose post-mastectomy pain syndrome after surgery in women with resectable breast cancer.

Secondary

* Determine the psychological and sociological factors that predispose post-surgical pain in these patients.
* Evaluate emotional distress over time in these patients.
* Evaluate the acute and chronic pain over time in these patients.

This is a multicenter study. Patients complete multiple questionnaires, including Hospital Anxiety and Depression Scale (HAD), Maudsley Personality Inventory (MPI), PCS, and QLQ-C30, to evaluate psychological variables (alexithymia, neurosis, repression of negative emotions, solicitude, dramatization, emotional distress) and quality of life.

Post-mastectomy chronic pain (PMCP) syndrome is measured immediately after surgery and at 24 hours, day 6, and 5 months post-surgery.

A subgroup of patients (20 with PMCP and 20 without PMCP) are followed at months 5 and 6 months post-surgery for medication use, pathological problems, morbid events, family history, and environmental factors.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Mastectomy or lumpectomy, including axillary lymph node dissection, planned
* Analgesic fixed (or ordered) the morning of surgery

  * No stage III analgesic planned
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* WHO performance status 0-2
* Other prior malignancy allowed
* No American Society of Anesthesiologists' class IV
* No contraindication or drug addiction
* No uncontrolled conditions, including any of the following:

  * Diabetes
  * Thyroid disease
  * Neuropsychiatric disease
  * Infection
  * Insufficient coronary function
  * NYHA class III-IV heart disease

PRIOR CONCURRENT THERAPY:

* No recent major surgery
* No participation in another medical or surgical clinical trial in the past 30 days
* Prior breast surgery for a benign lesion or malignant lesion allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Presence of post-mastectomy pain syndrome | At 3 months after surgery
  Pain is measured using a visual analog scale (VAS), ranging from 0 (no pain) to 100 (worst pain ever).
  A participant is considered to have pain syndrome if VAS score is >= 70.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Dixmerias, MD, Study Chair — Institut Bergonié

IPD SHARING:
Plan to Share IPD: No